CLINICAL TRIAL: NCT00827476
Title: Phase 1 Study to Improve Results of Human Ovarian Transplantation
Brief Title: Improving Human Ovarian Transplantation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Israel Science Foundation (Other)
Responsible Party: Ariel Revel, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0530-08-HMO- CTIL
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Fertility Preservation
Keywords: ovary; human; transplantaion; ovarian failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ovarian transplantation (Experimental): tissue will be used for xenotransplantation or in vitro culture
  Interventions: Procedure: ovarian transplantation

INTERVENTIONS:
Procedure: ovarian transplantation — ovarian xenotransplantation or in vitro culture

SUMMARY:
we will perform xenotransplantation and in vitro culture of ovarian tissue from patients undergoing ovarian cortex cryopreservation.

DETAILED DESCRIPTION:
Ovarian tissue is removed by laparoscopy and only in patients facing premature ovarian failure due to chemotherapy.Tissue for research will consist either of a small portion (<10%) of the cortex for preservation for young women. another source of ovarian tissue for research will be obtained following consent from family of patients who have died of the disease and have previously frozen ovarian tissue.

ELIGIBILITY:
Inclusion Criteria:

* tissue previously obtained

Exclusion Criteria:

* no tissue available or no consent

Ages: 5 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
improving folliculogenesis and oocuyte maturation after ovarian transplantation | 2 years